CLINICAL TRIAL: NCT06673069
Title: A Phase 1b Study to Assess the Safety, Tolerability, and Pharmacokinetics of ION269 in Adults With Down Syndrome (Hero Study)
Brief Title: Hero: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics (PK) and Pharmacodynamics (PD) of ION269 in Participants With Down Syndrome (DS) at Risk for Alzheimer's Disease (AD)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ION269-CS1; 2023-509257-31-00 (EU CTIS Number); U1111-1306-9498 (Other: WHO Number)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Alzheimer Disease; Down Syndrome
MeSH Terms: conditions — Alzheimer Disease; Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Participants will receive a single dose of ION269.
  Interventions: Drug: ION269
- Cohort 2 (Experimental): Participants will receive a single dose of ION269.
  Interventions: Drug: ION269
- Cohort 3 (Experimental): Participants will receive a single dose of ION269.
  Interventions: Drug: ION269

INTERVENTIONS:
Drug: ION269 — Administered as intrathecal (IT) injection.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of ION269 in adults with Down syndrome with evidence of brain amyloid positivity.

DETAILED DESCRIPTION:
This is a phase 1b multi-center, open-label, single ascending dose (SAD) study in adult participants with Down syndrome with evidence of brain amyloid positivity. Participants will be examined in 3 separate cohorts and will receive a single dose of study drug during the 36-week treatment period, followed by a 4-week follow-up period.

ELIGIBILITY:
Inclusion criteria:

1. Has a reliable study partner, that is, a parent, sibling, or caregiver ≥ 21 years of age, who has known the participant for > 6 months (i.e., a reliable and competent individual with a close relationship with the participant) and is capable of providing accurate information about the participant's history, can attend all scheduled study visits and provide feedback regarding the participant's symptoms and performance as described in the protocol, and can comply with all study requirements and activities.
2. Has a diagnosis of Down syndrome and has an intelligence quotient (IQ) ≥ 45.
3. Has evidence of amyloid pathology on amyloid-positron emission tomography (PET) scan.
4. Is assessed as being cognitively stable.
5. Is in good health as evidenced by medical history, physical, and neurological examination, and with no diagnosis of dementia or mild cognitive impairment.

Exclusion criteria:

1. Has unstable psychiatric illness, including psychosis, or untreated major depression within 90 days before Screening, as determined by the Investigator.
2. Has any unstable medical condition likely to hamper the evaluation of safety and/or efficacy of the Study Drug (e.g., moderate or severe untreated obstructive sleep apnea, medical history of clinically significant B12 or folate deficiency that is currently uncontrolled, clinically significant abnormalities of thyroid function, stroke, or other cerebrovascular conditions), as per Investigator's judgment.
3. Is unable to complete MRI and amyloid/tau-PET procedures or has any contraindications to having a brain MRI (e.g., MRI-incompatible pacemaker, aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed without requiring general anesthesia).

Note: Other protocol defined inclusion/exclusion criteria may apply.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2024-12-20 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to approximately Week 40
Number of Participants With Change from Baseline in Laboratory Assessments | Up to approximately Week 40
Number of Participants With Change from Baseline in Cerebrospinal fluid (CSF) Safety Laboratory Assessments | Up to approximately Week 40
Number of Participants With Change From Baseline in Vital Signs | Up to approximately Week 40
Number of Participants With Change From Baseline in Weight | Up to approximately Week 40
Number of Participants With Change From Baseline in Electrocardiogram (ECG) | Up to approximately Week 40
Number of Participants With Change From Baseline in Suicide Risk Measured by Columbia Suicide Severity Rating Scale [C-SSRS] Child Version | Up to approximately Week 40
Number of Participants With Change From Baseline in Physical and Neurological Examination Findings | Up to approximately Week 40

SECONDARY OUTCOMES:
CSF Concentrations of ION269 | Pre-dose and post-dose at multiple timepoints up to Week 40
Area Under the Plasma Concentration-time Curve (AUC) of ION269 From Time 0 to Time of Last Measurable Concentration | Pre-dose and post-dose at multiple timepoints up to Week 40
Maximum Observed Plasma Concentration (Cmax) of ION269 | Pre-dose and post-dose at multiple timepoints up to Week 40
Time to reach Cmax (Tmax) of ION269 | Pre-dose and post-dose at multiple timepoints up to Week 40
Change From Baseline in Concentration of CSF Soluble Amyloid Precursor Protein Alpha (sAPPα) | Baseline (Day 1) and Week 36
Change From Baseline in Concentration of CSF Soluble Amyloid Precursor Protein Beta (sAPPβ) | Baseline (Day 1) and Week 36

CONTACTS AND LOCATIONS:
Locations (6):
- United States (5):
  - Ionis Investigative Site, Indianapolis, Indiana
  - Ionis Investigative Site, Kansas City, Kansas
  - Ionis Investigative Site, Lexington, Kentucky
  - Ionis Investigative Site, St Louis, Missouri
  - Ionis Investigative Site, Madison, Wisconsin
- Ionis Investigative Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Ionis may share anonymized individual participant data, aggregated clinical data, and other types of data that support the results in this study. Data requests from qualified researchers will be considered once all three of the following criteria are met: (1) 12 months from marketing approval of the study drug in both the United States and European Union; (2) 18 months from conclusion of the study; and (3) 6 months from publication of study article. Access would be via a secure environment and is contingent upon approval of a research proposal and entry into an appropriate data use agreement. Requests to access data can be submitted via the website https://vivli.org/ourmember/ionis/.